CLINICAL TRIAL: NCT07104812
Title: Impact of 1 mg Osilodrostat Therapy on Mild Autonomous Cortisol Secretion (MACS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Principal Investigator, Irina Bancos, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-007009
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mild Autonomous Cortisol Secretion; Autonomous Cortisol Secretion (ACS)
Keywords: hypercortisolism; cortisol excess; Adrenal adenoma; Adrenal hyperplasia; Cushing Syndrome
MeSH Terms: conditions — Cushing Syndrome; ACTH Syndrome, Ectopic; Adrenal Hyperplasia, Congenital | interventions — Osilodrostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mild autonomous cortisol secretion (MACS) (Experimental): Women and men diagnosed with MACS who are patients at Mayo Clinic.
  Interventions: Drug: Osilodrostat 1 MG

INTERVENTIONS:
Drug: Osilodrostat 1 MG — Osilodrostat 1 mg administered between noon and 6 pm daily, for 4 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of 1 mg osilodrostat therapy in patients with mild autonomous cortisol secretion (MACS), and to determine the impact on 24h urine steroid metabolome and circadian cortisol/cortisone concentrations

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age ≥ 18 years
* Diagnosed with MACS

  * At least 2 abnormal post-dexamethasone cortisol results:

    i. 1 mg post-dexamethasone cortisol >1.8 mcg/dL or ii. 8 mg post-dexamethasone cortisol >1 mcg/dL
  * Historical dexamethasone suppression test results can be used if performed within 24 months prior to enrollment.
* Adrenal imaging phenotype consistent with benign disease (adrenal adenoma/s, macronodular or micronodular adrenal hyperplasia)
* At least one of the following comorbidities:

  * Obesity (BMI>30 kg/m2)
  * Dysglycemia
  * Dyslipidemia
  * Hypertension
  * Osteopenia
  * Osteoporosis
  * Fragility fractures
* Ability to take oral medication and be willing to adhere to the study intervention regimen
* For persons of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of ≤ 5% per year during the treatment period and for 1 month after the last dose of study treatment.

Exclusion Criteria:

* Planned alternative therapy for MACS during the study period
* Current use of oral exogenous glucocorticoid therapy
* Current use of opioid therapy >20 MME/day
* Planned use of oral exogenous glucocorticoid therapy
* Planned use of opioid therapy >20 MME/day
* Use of injectable glucocorticoid within the last 6 weeks or anticipated glucocorticoid use during the study period.
* Hypokalemia of hypomagnesemia at baseline visit
* Prolonged QTc on baseline ECG
* Concomitant therapy with medications likely to lead to drug-drug interactions (based on PI review).
* Investigator's judgement based on history/physical examination that a comorbidity or concomitant medication may impact the hypothalamic-pituitary-adrenal axis or steroid metabolome
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnancy or lactation
* Known allergic reactions to osilodrostat
* Suspected false positive post-dexamethasone cortisol results due to increased metabolism, poor absorption, or noncompliance with dexamethasone.
* Treatment with another investigational drug or other intervention within lower than specific therapy washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 4 weeks
  Number of adverse events
Adrenal insufficiency | 4 weeks
  Number of subjects to experience adrenal insufficiency, defined as combined measurements of cortisol < 7 mcg/dL and ACTH>60 pg/dL or single cortisol < 5 mcg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Irina Bancos, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No